CLINICAL TRIAL: NCT03416309
Title: Personalization of AntiTB Treatment: Evaluation of Pharmacological Determinants of Treatment Response
Acronym: PAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Collaborators: Research Center Borstel (Other)
Responsible Party: Principal Investigator, Ilaria Motta, Principal Investigator, University of Turin, Italy
Other Study IDs: PAT_Study
Record Dates: First submitted 2018-01-10; First posted 2018-01-31 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Tuberculosis, Pulmonary
Keywords: pharmacokinetics; pharmacogenetics; Time To Positivity
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — DNA samples will be stored in an appropriate place recognizable by inscriptions or encodings that will in any way be attributable to any personal or sensitive data of the patient in full respect of privacy, and will be accessible only by the staff involved in the study in full compliance with the safety standards.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate the possible correlation of plasma drug concentrations with Time To Positivity (TTP) in liquid culture in patients with active pulmonary multi sensitive TB in the first two weeks of treatment. Secondary aims are: the correlation between plasma drug concentrations and hepato/neuro toxicity; the impact of different allelic variants on PK data, toxicity and TTP in liquid culture; the feasibility of using dried blood/plasma spots to measure plasma concentrations of anti-TB drugs and determine genetic polymorphisms.

DETAILED DESCRIPTION:
A longitudinal observational multicentred study will be conducted in patients with diagnosis of active pulmonary TB.

The following variables will be recorded:

* demographic variables: age, gender, ethnicity, SNPs for NAT2, SLCO1B1, ABCB1 and VDR;
* clinical variables: weight, height, renal function tests, liver function tests, vitamin D (25-OH vitamin D) level, albuminemia, serology for HIV, HCV, presence of comorbidities (e.g. diabetes mellitus), visual acuity test, presence of neuropathic symptoms;
* microbiological variables: phenotypic and genotypic drug sensitivity test results, sputum Mycobacterium tuberculosis DNA (PCR), microscopy, culture, Time To Positivity (TTP) in liquid culture, IGRA test (if performed), history of previous treatments, location of pulmonary lesions, presence of extra-pulmonary locations;
* therapeutic variables: start/end of treatment, treatment interruptions, dose mg/kg, route of administration.

The patients will received standard antitubercular drugs according to international guidelines (RIF 10 mg/kg, INH 5 mg/kg maximum dose 300 mg, ETB 15-20 mg/kg, PZA 25 mg/kg maximum dose 2000 mg) in fasten condition, once daily.

To measure plasma concentrations four blood samples (Lithium heparin 7 ml tubes) will be collected at 0, 2, 4 and 6 hours post dose. This analysis will be performed at 7 and 14 days after the beginning of anti-TB treatment.

For the pharmacogenetic analysis a blood sample (EDTA 4 ml tube) will be collected at the baseline.

Sputum samples will be collected at baseline, 7 and 14 days for Mycobacterial culture.

Medical visits and blood samples (for LFTs) will be performed at baseline, 7 and 14 days to investigate neuro and hepato- toxicity.

Pharmacokinetics After the collection the samples will be centrifugated (3000 rev min-1 at 4°C for 10 min) and plasma will be frozen at - 20°C in 2 aliquots (1 mL of volume) and will be delivered to the Laboratory of Pharmacokinetics and Pharmacogenetics of the University of Torino Amedeo di Savoia Hospital, ASLTO2, Torino, Italy.

Plasma concentrations of all four drugs will be measured using liquid chromatography coupled with tandem mass-spectroscopy (allowing high sensitivity despite small sample volumes). Collected concentration-time data will be evaluated by a non-compartmental approach to characterize the pharmacokinetic properties at steady-state. AUC, maximum (Cmax) and minimum (Cmin) drug levels and plasma elimination half-life will be used to assess the enzymatic induction properties of these drugs. Pharmacogenomics (PG) DNA will be extracted from whole blood using QIamp DNA Mini Kit (Quiagen, Valencia, CA). Purified and eluted DNA will be directly used for real-time PCR (BIORAD, Milano, Italia) reaction. The allelic discrimination analysis will be performed using the TaqMan assays (Applied Biosystems, Foster City, CA).

Analyzed SNPs will be:

ABCB1 3435C>T (rs1045642), OATP1B1 521T>C (rs4149056) e OATP1B1 85-7793T>C (rs4149032), PXR 63396C>T (rs2472677), BsmI G>A (rs1544410).

and NAT2 G>A (rs1799930). Dried blood spots (DBSs) and Dried plasma spots (DPSs) Method for the determination of plasma concentrations on DPSs will be developed and validated by our laboratory. In the study, the blood samples for evaluation on DPSs will be obtained only from subjects of our institute. After centrifugation (3000 rev min-1 at 4°C for 10 min) 100 μ l plasma will be spotted onto each glass filter (purchased from Laboratori Biomicron srl, Italy) and used for pharmacokinetic (PK) analysis. The remaining plasma will be used as controls in the analysis.

For the pharmacogenetic (PG) analysis venous blood samples will be obtained from all subjects and whole blood (50 μ l per spot) will be spotted on DBS Whatman 903 protein saver cards (VWR International, Milan, Italy).

DBS will be inserted in a foil bag with desiccant (Foil Bag and Desiccant Packs, purchased from Laboratori Biomicron srl, Italy) and then stored at room temperature. After a maximum of 30 days samples will be delivered to the Laboratory of Pharmacokinetics and Pharmacogenetics of the University of Torino Amedeo di Savoia Hospital, ASLTO2, Torino, Italy. They will be stored at - 20°C until analysis will be performed (within 3 months from collection).

Time To Positivity Time to positivity on sputum cultures at baseline, 7 and 14 days will be calculated using software BD Epicenter integrated in BACTEC MGIT System (Mycobacteria Growth Indication Tube) 960. Default time is 42 days.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* age >=18 years;
* pulmonary tuberculosis defined by positive sputum microscopy (waiting for culture confirmation)
* sensitivity to first-line anti-TB drugs;
* normal liver and renal function.

Exclusion Criteria:

* severe malnutrition;
* HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pulmonary TB referred from other primary health centers All the patients with diagnosis of pulmonary DS (drug sensitive) TB will be enrolled.
  The patients will received standard antitubercular drugs according to international guidelines (RIF 10 mg/kg, INH 5 mg/kg maximum dose 300 mg, ETB 15-20 mg/kg, PZA 25 mg/kg maximum dose 2000 mg) in fasten condition, once daily.
Sampling Method: Probability Sample
Enrollment: 257 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Correlation between AUC of RHZE and TTP | 1 week from start of treatment
  Investigate the correlation of plasma drug concentrations (Rifampicin, Isoniazid, Ethambutol and Pyrazinamide, HRZE) with the change in Time To Positivity (TTP) in liquid culture in patients with active pulmonary TB between the baseline and the first week of treatment.
Correlation between AUC of RHZE and TTP | 2 weeks from start of treatment
  Investigate the correlation of plasma drug concentrations (Rifampicin, Isoniazid, Ethambutol and Pyrazinamide, HRZE) with the change in Time To Positivity (TTP) in liquid culture in patients with active pulmonary TB between the baseline and the second week of treatment.

SECONDARY OUTCOMES:
Correlation between AUC of RHZE and toxicity | 1 week and 2 weeks from start of treatment
  Investigate the correlation of plasma drug concentrations (Rifampicin, Isoniazid, Ethambutol and Pyrazinamide, HRZE) with hepatotoxicity (increase of AST and/or ALT) and neurotoxicity (peripheral neuropathy)
Correlation between PG and AUC of RHZE | 1 week and 2 weeks from start of treatment
  Investigate the impact of different allelic variants of NAT2, SLCO1B1, ABCB1, VDR on AUC of RHZE toxicity and TTP in liquid culture
Assess the consistency of results using of DPS for measuring the plasma drug concentrations | 1 week and 2 weeks from start of treatment
  Assess the consistency of using dried plasma spots to measure plasma concentrations of anti-TB drugs comparing to plasma samples
Correlate AUC of RHZE with antiTB response | 6 months after end of treatment
  A pharmacometric model will be develop to correlate pharmacokinetics (AUC of RHZE) with the anti-TB treatment response (clinical and TTP) of the standard first-line anti-TB regimen.
Correlate PG with antiTB response | 6 months after end of treatment
  A pharmacometric model will be develop to correlate PG with the anti-TB treatment response (clinical and TTP) of the standard first-line anti-TB regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Motta, MD, Principal Investigator — University of Turin, Italy
Locations (1):
- Ospedale Amedeo di Savoia, Torino, Italy

IPD SHARING:
Plan to Share IPD: Undecided
We can share anonymous data upon request